CLINICAL TRIAL: NCT00005409
Title: Longitudinal Studies of Blood Pressure in the Elderly
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4327; R03HL046923 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To study further the association between blood pressure mortality among those who participated in both the Hypertension Detection and Follow-up Program (HDFP) screen and the East Boston Established Populations for Epidemiologic Studies in the Elderly (EPESE) study.

DETAILED DESCRIPTION:
BACKGROUND:

In middle-age, level of blood pressure (BP) is a strong and independent predictor of both total and cardiovascular disease (CVD) mortality. However, among the elderly, recent short-term observational studies, including the East Boston Established Populations for Epidemiologic Studies in the Elderly (EPESE), have raised the possibility of a J-shaped curve. In a study of short-term mortality, low blood pressures were positively associated with total and cardiovascular disease mortality. However, a further analysis confined to the 2079 (68 percent) of this cohort who were also screened nine years previously for the Hypertension Detection and Follow-Up Program showed the more conventional positive linear relationship between systolic blood pressure, and no association between diastolic blood pressure and mortality. The observations of higher short-term total and cardiovascular disease mortality at lower blood pressure levels among the elderly could have reflected a particular susceptibility to deleterious consequences of drug therapy for high blood pressure. Alternatively, such a finding might have been artifactual, due to survival bias or confounding by co-morbid conditions.

DESIGN NARRATIVE:

Linking data from the HDFP and the EPESE studies, the investigators examined change in blood pressure, antihypertensive medication use, and mortality over a 15-year period. With regard to the association between lower blood pressure and increased mortality, they determined whether the relationship previously observed reflected a fall from normotensive levels as opposed to a consistently low blood pressure. With regard to the upper end of the mortality curve, they assessed the effect of antihypertensive drug treatment on mortality as compared to those with untreated hypertension. The latter question had particular public health significance because questions remained about the risk-to-benefit ratio of antihypertensive drug treatment in this age group. Furthermore, they also described changes in blood pressure in this population and medication usage patterns over time and correlated type of medication and mortality.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-05; Study Completion 1993-04 (Actual)

REFERENCES:
- [Background] Glynn RJ, Field TS, Satterfield S, Hebert PR, Buring JE, Taylor JO, Hennekens CH. Modification of increasing systolic blood pressure in the elderly during the 1980s. Am J Epidemiol. 1993 Sep 15;138(6):365-79. doi: 10.1093/oxfordjournals.aje.a116869. PMID 8213742